CLINICAL TRIAL: NCT01684852
Title: Non Interventional Study to Evaluate the Efficacy and Tolerability of Ectoin Containing Ophthalmic Solution (BAT04) Compared to HA Eye Drops in the Treatment of Dry Eye Disease
Brief Title: Non Interventional Study to Evaluate the Efficacy and Tolerability of Ectoin Containing Ophthalmic Solution
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: PPL-046; NIS BAT04
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye, sicca, HA, Hyaluronic Acid, ectoin, ectoine, bitop
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medical device, drug-like

SUMMARY:
This is a comparative, open label, parallel group, non interventional study to further demonstrate the efficacy and tolerability of BAT04. In addition the efficacy and safety shall be compared to Hyaluronic acid (HA)-Product. The patient applies BAT04 or HA-Product according to the instructions for use six times daily in both eyes over a period of 28 days. Response to treatment is recorded at day 28.

ELIGIBILITY:
Inclusion Criteria:

* Male or female person aged 18 years
* Demonstrated mild to moderate keratoconjunctivitis sicca ( "dry eye")
* Acute symptoms of dry eye: DEWS 1-3
* tear break-up time TBUT <10s
* agreement to abide by the routinely provided doctor's appointment for follow-up (reflected in the planned visits of observation plan resist)

Exclusion Criteria:

* inflammation of the anterior segment or trauma
* Contact lens wearers
* Any disease that can, in the opinion of the treating physician to affect the outcome of the study.
* Patients with known intolerance to one of the substances used
* Surgical procedures to the eyes in the last 6 weeks before inclusion in the trial
* patients with addictive disorders or substance abuse fallow in the past 12 months, as well as persons incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic The selection of appropriate patients for the observational study is made by the individual physician in his treatment decisions in consultation with the individual patient
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tear Break Up Time | V1 and V2

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Messmer, MD, Principal Investigator — Augenklinik der LMU Klinikum der Universität München
Locations (5):
- Germany (5):
  - Dr. Peter Otto, Bad Liebenwerda
  - Dr. Insa Beddermann, Duderstadt
  - Augenklinik mit Poliklinik, Erlangen
  - Augenklinik der LMU Klinikum der Universität Muenchen, München
  - Augenabteilung am St. Franziskus-Hospital Münster, Münster